CLINICAL TRIAL: NCT00911482
Title: FFA Production From Triglyceride-Rich Lipoproteins
Brief Title: Production of Free Fatty Acids From Blood Triglycerides
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: John M. Miles, MD, Mayo Foundation
Other Study IDs: 08-001493; R01HL067933 (NIH)
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance; Dyslipidemias
Keywords: Type 2 Diabetes; Dyslipidemia; FFA; Triglycerides; Tracers
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Dyslipidemias

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma samples obtained during the study are stored for lipid analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Diabetes/weight loss: 12 individuals with type 2 diabetes and hypertriglyceridemia
- Nondiabetic/hypertriglyceridemic: 10 insulin resistant nondiabetic individuals with dyslipidemia
- Normotensive/nondiabetic: 10 insulin resistant, normotensive, nondiabetic individuals
- Insulin resistant/dyslipidemic: 14 insulin resistant nondiabetic individuals with dyslipidemia

SUMMARY:
The overall hypothesis of these studies is that circulating triglycerides, coming primarily from fat in the diet, are an important source of free fatty acids. Free fatty acids are the major fat fuel in the body, and when they are elevated in the blood they are thought to raise the risk of cardiovascular disease by causing insulin resistance (in some cases leading to diabetes), raising blood pressure, and other effects. The investigator will use sophisticated methods for tracing triglycerides and free fatty acids in the blood. These methods involve the administration of low doses of radioactive and stable isotopes of naturally occurring fats. The studies will determine the contribution of triglycerides to free fatty acids in normal people and also in people with diabetes.

DETAILED DESCRIPTION:
Lipid energy is transported in the blood in several forms, including chylomicrons and free fatty acids (FFA). Chylomicrons are key elements in the absorption and storage of dietary fat, and also play a role in the pathogenesis of atherosclerosis via the production of remnant particles, but their role as a direct fuel source has not been explored. FFA are the major lipid fuel in the body, and increases in their concentration have been shown to cause insulin resistance, endothelial dysfunction and increases in the production of very low density lipoproteins. FFA are released into the blood through the action of hormone sensitive lipase on triglyceride stores in fat cells. Very little is known about the role of chylomicrons in FFA metabolism, but the potential contribution of chylomicrons to FFA is considerable, especially in people who consume high fat diets. Initial studies indicate that in addition to the role of chylomicrons in fat storage, a portion of chylomicron fatty acids are released as FFA in a process called "spillover". These studies indicate that the contribution of chylomicrons to FFA is increased in type 2 diabetes. A study of spillover in the splanchnic bed found very high rates of splanchnic spillover in overweight and obese individuals with hypertriglyceridemia. Extremely accurate and precise methods have been developed by the investigator for the measurement of the concentration and specific activity of FFA and chylomicron triglyceride fatty acids in plasma. In addition, a tracer method for accurately determining the kinetics of chylomicrons has been developed. In the proposed studies, the tracer technique will be used to systematically investigate the contribution of chylomicrons to total FFA availability. The technique will be applied to normal subjects at rest and after exercise, as well as subjects with type 2 diabetes mellitus and hypertriglyceridemia. Specifically, these studies will: 1) determine whether weight loss in people with type 2 diabetes reduces spillover from chylomicrons; 2) determine whether acute lowering of FFA with insulin infusion reduces spillover in nondiabetic individuals with dyslipidemia; 3) determine whether noninsulin-mediated lowering of FFA reduces spillover in diabetic individuals with dyslipidemia, and 4) determine whether obese, insulin-resistant individuals have increased spillover in the splanchnic bed.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Atherogenic dyslipidemia
* Obesity

Exclusion Criteria:

* Kidney disease
* Liver disease
* Coronary artery disease
* Retinopathy
* Neuropathy

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers from the region around Rochester, Minnesota who meet the inclusion criteria will be recruited.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Spillover of free fatty acids from chylomicrons | Measured at 1 to 6 days

CONTACTS AND LOCATIONS:
Overall Officials: John M. Miles, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States